CLINICAL TRIAL: NCT01547377
Title: Effect of Zinc and Selenium Supplementation in Patients With Atherosclerosis Treated With Statins
Brief Title: Zinc and Selenium Supplementation in Atherosclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Karine C M Sena-Evangelista, Principal Investigator, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PROJ-981-199697778
Record Dates: First submitted 2012-02-22; First posted 2012-03-07 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Dietary Selenium Deficiency; Dietary Zinc Deficiency
Keywords: atherosclerosis; zinc and selenium status; rosuvastatin; oxidative stress biomarkers; inflammation biomarkers
MeSH Terms: conditions — Atherosclerosis | interventions — Zinc; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- zinc and selenium supplementation (Experimental): Patients received 10 mg rosuvastatin, concomitantly with zinc (30mg/d) and selenium (150μg/d) supplementation during 4 months
  Interventions: Dietary Supplement: zinc and selenium supplementation
- rosuvastatin + placebo (Placebo Comparator): Patients received 10 mg rosuvastatin concomitantly placebo pills similar zinc and selenium supplementation
  Interventions: Other: rosuvastatin + placebo

INTERVENTIONS:
Dietary Supplement: zinc and selenium supplementation — Data from patients were obtained at beginning and after four months of treatment with 10 mg rosuvastatin, concomitantly with zinc (30mg/d) and selenium (150μg/d) supplementation or placebo. The anthropometric and dietary data, zinc and selenium concentrations in plasma and erythrocyte, lipid profile, electronegative LDL (LDL(-)), anti- electronegative LDL, Ac-LDL(-) immune complexes, GPx and SOD activities, IL-6 and hs-CRP were evaluated in all patients
  Other Names: Zinc and selenium supplementation + rosuvastatin
  Arms: zinc and selenium supplementation
Other: rosuvastatin + placebo — Data from patients were obtained at beginning and after four months of treatment with 10 mg rosuvastatin, concomitantly with zinc (30mg/d) and selenium (150μg/d) supplementation or placebo. The anthropometric and dietary data, zinc and selenium concentrations in plasma and erythrocyte, lipid profile, electronegative LDL (LDL(-)), anti- electronegative LDL, Ac-LDL(-) immune complexes, GPx and SOD activities, IL-6 and hs-CRP were evaluated in all patients
  Other Names: placebo group
  Arms: rosuvastatin + placebo

SUMMARY:
The aim of this randomized double-blind study was to evaluate the effect of oral zinc and selenium supplementation on oxidative stress and inflammation biomarkers as well as the status of zinc and selenium in patients with atherosclerosis and angina stable treated with rosuvastatin. The hypotheses tested in this study were: Treatment with rosuvastatin impairs zinc and selenium status in patients with atherosclerosis and stable angina? Zinc and selenium supplementation, concomitantly with rosuvastatin, influences the antioxidant and anti-inflammatory as well as the status of minerals?

DETAILED DESCRIPTION:
The study included 47 men and 29 women, average age around 60 years, with coronary atherosclerosis diagnosed by angiography. Data from patients were obtained at beginning and after four months of treatment with 10 mg rosuvastatin, concomitantly with zinc (30mg/d) and selenium (150μg/d) supplementation or placebo. The anthropometric and dietary data, zinc and selenium concentrations in plasma and erythrocyte, lipid profile, electronegative LDL (LDL(-)), anti- electronegative LDL, Ac-LDL(-) immune complexes, GPx and SOD activities, IL-6 and hs-CRP were evaluated in all patients.

ELIGIBILITY:
Inclusion Criteria:

* The study included adult and elderly patients, with coronary atherosclerosis and stable angina diagnosed by angiography showing ≥ 70% stenosis of the vessel lumen in at least one segment of a major epicardial artery or ≥ 50% stenosis of the diameter of the left main coronary artery, stable angina

Exclusion Criteria:

* Cardiac complications or other serious diseases such as:

  * thyroid,
  * hematologic,
  * congenital,
* autoimmune liver disease,
* kidney failure,
* cancer,
* associated infections,
* osteoporosis,
* post-operative,
* use of:

  * antacids,
  * antibiotics and
  * vitamin-mineral supplements,
* alcohol and
* current smoking.

Ages: 41 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2008-01; Primary Completion 2009-04 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in zinc and selenium status at 4 months | Baseline and 4 months
  We evaluated the effects of 10mg rosuvastatin treatment as well as the effect of treatment with 10 mg rosuvastatin, concomitantly with zinc (30mg/d) and selenium (150μg/d) supplementation on plasma zinc and selenium and on erythrocyte zinc and selenium.

SECONDARY OUTCOMES:
Change from baseline in lipid profile at 4 months | Baseline and 4 months
  We evaluated the effects of 10mg rosuvastatin treatment as well as the effect of treatment with 10 mg rosuvastatin, concomitantly with zinc (30mg/d) and selenium (150μg/d) supplementation on total cholesterol, LDL, non-HDL cholesterol and, triglycerides.
Change from baseline in zinc and selenium status at 4 months | Baseline and 4 months
  We evaluated the effects of 10mg rosuvastatin treatment as well as the effect of treatment with 10 mg rosuvastatin, concomitantly with zinc (30mg/d) and selenium (150μg/d) supplementation on LDL (-), anti-LDL (-), immune complexes concentrations, SOD and GPx activities.
Change from baseline in inflammation biomarkers status at 4 months | Baseline and 4 months
  We evaluated the effect of oral zinc and selenium supplementation, concomitant with rosuvastatin treatment, on hs-CRP and IL-6 levels.

CONTACTS AND LOCATIONS:
Overall Officials: Dulcineia SP Abdalla, PhD, Study Director — University of Sao Paulo; Lucia FC Pedrosa, PhD, Study Director — University of Rio Grande do Norte
Locations (1):
- Onofre Lopes University Hospital, Natal, Rio Grande do Norte, Brazil

REFERENCES:
- [Derived] Sena-Evangelista KC, Pedrosa LF, Paiva MS, Dias PC, Ferreira DQ, Cozzolino SM, Faulin TE, Abdalla DS. The hypolipidemic and pleiotropic effects of rosuvastatin are not enhanced by its association with zinc and selenium supplementation in coronary artery disease patients: a double blind randomized controlled study. PLoS One. 2015 Mar 18;10(3):e0119830. doi: 10.1371/journal.pone.0119830. eCollection 2015. PMID 25785441